CLINICAL TRIAL: NCT04180462
Title: Randomized Controlled Trial to Evaluate an Implementation Strategy to Increase Optimal Use of HPV Vaccine in Primary Care
Brief Title: Increasing Optimal Use of HPV Vaccination in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 201911030; 1R01CA235615-01A1 (NIH)
Record Dates: First submitted 2019-11-26; First posted 2019-11-27 (Actual); Results first posted 2024-02-20 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Human Papillomavirus Vaccines
Keywords: Implementation Strategy; Quality Improvement
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Practices randomly assigned to this arm will receive the multi-component intervention.
  Interventions: Other: Practice Facilitation; Other: Education; Other: Audit and Feedback; Other: Communication Strategy
- Wait list control group (No Intervention): Practices randomly assigned to this arm will be offered the intervention in the last two years of the study.

INTERVENTIONS:
Other: Practice Facilitation — Practice facilitation to support quality improvement methods to effect practice change to develop a sustainable HPV vaccine delivery system.
  Arms: Intervention Group
Other: Education — An educational video to increase the provider's knowledge about guideline recommendations and patient and practice benefits of vaccination by age 13.
  Arms: Intervention Group
Other: Audit and Feedback — Audit and feedback of vaccine coverage to increase motivation to engage in practice change.
  Arms: Intervention Group
Other: Communication Strategy — A communication strategy to improve the provider's communication skills and their self-efficacy to address parental hesitation.
  Arms: Intervention Group

SUMMARY:
Washington University will evaluate the effectiveness of a multi-component implementation strategy to increase use of HPV vaccine in primary care practices.

DETAILED DESCRIPTION:
The investigators at Washington University will complete a cluster-randomized trial to evaluate the effectiveness of a multi-component implementation strategy (the intervention) to increase use of the HPV vaccine according to CDC guidelines. The unit of randomization is a community-based, primary care pediatric practice. Twenty practices will be randomized into two groups, the intervention group (n=10) or a wait-list control group (n=10). The intervention will be implemented over 2-years and includes: 1) an educational video for providers; 2) audit and feedback of vaccine coverage; 3) a communication strategy; and 4) practice facilitation.

The primary outcome of HPV vaccination by age 13 will be assessed at 24 months, and at 36 months to assess if change is sustained.

ELIGIBILITY:
Inclusion Criteria

Practices:

* Community-based pediatric primary care practices with 2 or more providers.
* Providers who deliver wellness care to preteens and adolescents.
* Willingness to participate in the practice facilitator-guided QI process.

Providers:

* Providers who deliver wellness care to preteens and adolescents.
* Willingness to complete study questionnaires.
* Willingness to participate in the practice facilitator-guided QI process.

EXCLUSION CRITERIA

* Practices and providers may be excluded at the discretion of the PI.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2024-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allison King, M.D., Ph.D., MPH, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu
- See also: Washington University: Pediatric & Adolescent Ambulatory Research Consortium — https://paarc.wustl.edu/

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: practices
Period: Overall Study
Arm/Group | Intervention Group | Wait List Control Group
Started | 4362; 10 practices | 3025; 10 practices
24 Months Post-randomization | 2151; 10 practices (The 24 month post-randomization time point contains data collected from an individual set of pre-teen subjects and these subjects are not included in the 36 month post-randomization time point.) | 1615; 10 practices (The 24 month post-randomization time point contains data collected from an individual set of pre-teen subjects and these subjects are not included in the 36 month post-randomization time point.)
36 Months Post-randomization | 2211; 10 practices (The 36 month post-randomization time point contains data collected from an individual set of pre-teen subjects and these subjects are not included in the 24 month post-randomization time point.) | 1410; 9 practices (The 36 month post-randomization time point contains data collected from an individual set of pre-teen subjects and these subjects are not included in the 24 month post-randomization time point.)
Completed | 4362; 10 practices | 3025; 9 practices (One practice did not have data available for the 36 month post-randomization time point.)
Not Completed | 0; 0 practices | 0; 1 practices

BASELINE CHARACTERISTICS:
Groups:
- Intervention Group (24 Months Post-randomization); Intervention Group (36 Months Post-randomization): Practices randomly assigned to this arm will receive the multi-component intervention.
- Wait List Control Group (24 Months Post-randomization); Wait List Control Group (36 Months Post-randomization): Practices randomly assigned to this arm will be offered the intervention in the last two years of the study.
- Total: Total of all reporting groups
Arm/Group | Intervention Group (24 Months Post-randomization) | Wait List Control Group (24 Months Post-randomization) | Intervention Group (36 Months Post-randomization) | Wait List Control Group (36 Months Post-randomization) | Total
Number analyzed (Participants) | 2151 | 1615 | 2211 | 1410 | 7387
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2151 | 1615 | 2211 | 1410 | 7387
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 1037 | 818 | 1108 | 701 | 3664
  Male | 1113 | 797 | 1103 | 704 | 3717
  Unknown | 1 | 0 | 0 | 5 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 63 | 32 | 23 | 150
  Not Hispanic or Latino | 1634 | 1226 | 1692 | 1128 | 5680
  Unknown or Not Reported | 485 | 326 | 487 | 259 | 1557
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2 | 2 | 6
  Asian | 60 | 19 | 40 | 25 | 144
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 3 | 1 | 5
  Black or African American | 92 | 446 | 120 | 384 | 1042
  White | 1514 | 890 | 1560 | 819 | 4783
  More than one race | 30 | 45 | 15 | 35 | 125
  Unknown or Not Reported | 454 | 213 | 471 | 144 | 1282
Region of Enrollment [Number; unit: participants]
  United States | 2151 | 1615 | 2211 | 1410 | 7387

OUTCOME MEASURES:

1. Primary Outcome: Initiation of the HPV Vaccine 2-dose Series.
Description: The proportion of eligible preteens who initiate the HPV vaccine before their 13th birthday, at 24 months, post randomization
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Wait List Control Group
Number analyzed (Participants) | 2151 | 1615
Participants | 1723 | 1219

2. Primary Outcome: Completion of the HPV Vaccine 2-dose Series.
Description: The proportion of eligible preteens who complete the HPV vaccine before their 13th birthday, at 24 months, post randomization.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Wait List Control Group
Number analyzed (Participants) | 2151 | 1615
Participants | 1135 | 809

3. Secondary Outcome: Sustainability of the Intervention Benefit for Initiation of the HPV Vaccine.
Description: The proportion of eligible preteens who receive the 1st dose of HPV vaccine before their 13th birthday at 36 months, post randomization
Time Frame: 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Wait List Control Group
Number analyzed (Participants) | 2211 | 1410
Participants | 1812 | 1052

4. Secondary Outcome: Sustainability of the Intervention Benefit for Completion of the HPV Vaccine.
Description: The proportion of eligible preteens who complete the HPV vaccine before their 13th birthday, at 36 months, post randomization
Time Frame: 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Wait List Control Group
Number analyzed (Participants) | 2211 | 1410
Participants | 1279 | 703

ADVERSE EVENTS:
Time Frame: The only potential adverse event is breach of confidentiality. Regular monitoring will occur while the participants are on follow-up (up to 36 months)
Groups:
- Intervention Group (36 Month Post-randomization): Practices randomly assigned to this arm will receive the multi-component intervention.
Arm/Group | Intervention Group (24 Months Post-randomization) | Wait List Control Group (24 Months Post-randomization) | Intervention Group (36 Month Post-randomization) | Wait List Control Group (36 Months Post-randomization)
All-Cause Mortality (participants affected / at risk) | 0/2151 | 0/1615 | 0/2211 | 0/1410
Serious Adverse Events (participants affected / at risk) | 0/2151 | 0/1615 | 0/2211 | 0/1410
Other Adverse Events (participants affected / at risk) | 0/2151 | 0/1615 | 0/2211 | 0/1410

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-06): https://cdn.clinicaltrials.gov/large-docs/62/NCT04180462/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-16): https://cdn.clinicaltrials.gov/large-docs/62/NCT04180462/ICF_001.pdf